CLINICAL TRIAL: NCT00208884
Title: Terminal Graft Failure: A Combined Pathologic and Clinical Study
Brief Title: Terminal Graft Failure
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: 1001-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Orthotopic Heart Transplantation; Graft Failure
Keywords: pediatric; orthotopic heart transplantation; graft failure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
One of the risks associated with heart transplantation is failure of the graft. A graft is where the new heart is attached to the original vessels in the body. Approximately 10% of children suffer graft failure which, leads to heart failure and possible death. The problem is that we do not know some of the causes of graft failure thus, it is difficult to diagnose early and treat. Due to graft failure, lots of children are placed back on the transplant list and receive another new heart.

In this study, we plan to perform a retrospective chart review looking to see if we can correlate graft failure with a problem with the vessels called coronary allograft vasculopathy or rejection. In order to do this, we will collect data from patient's charts that have been diagnosed with graft failure and compare their clinical presentation/data to pathology reports of the explanted hearts from these children. Explanted hearts are the old transplanted hearts that are removed in order to put a new heart into the body. Explanted hearts at our institution are always sent to pathology for analysis thus it will be quite easy to perform this review.

DETAILED DESCRIPTION:
The objectives are to describe the pathology findings from the examination of the explanted heart and correlate them with clinical variables such as catheterization data.

Children's Healthcare of Atlanta performs approximately 12-15 heart transplants a year. To date, there have been 19 re-transplantations for late graft failure at Children's. The pathologic and clinical records of these 19 patients will be studied. All data collected will be entered into a database for future analysis.

Data Collection

A retrospective review of standard pathology findings from the examination of the explanted hearts will be conducted in order to determine the following:

1. Evidence of CAV (coronary allograft vasculopathy)
2. Evidence of Endocardial fibroelastosis
3. Evidence of Rejection (acute and chronic)
4. Evidence of Myocardial infarction
5. Evidence of Fibrosis
6. Evidence of Fatty infiltration

A retrospective review of patient charts will also be utilized to compare the pathologic findings to clinical data obtained prior to re-transplantation. The following information will be collected:

1. Type of transplant method
2. Patient age at time of transplant
3. Echocardiographic Data including Tissue Doppler Imaging (if available)
4. Catheterization data

   1. CAV as identified by coronary angiography
   2. Ventricular end-diastolic pressure
   3. Cardiac index
   4. Ventricular ejection fraction
5. Clinical rejection history

ELIGIBILITY:
Inclusion Criteria:

* retransplanted at Children's Healthcare of Atlanta for late graft failure

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19
Dates: Start 2003-10; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States